CLINICAL TRIAL: NCT00068042
Title: A Study To Compare The Efficacy And Safety Of Pegvisomant To That Of Sandostatin Lar Depot In Patients With Acromegaly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEGA-0435-003; A6291004
Record Dates: First submitted 2003-09-04; First posted 2003-09-08 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

INTERVENTIONS:
Drug: Pegvisomant
Drug: Sandostatin LAR

SUMMARY:
The purpose of the study is to determine if Pegvisomant is more efficacious than Sandostatin LAR Depot in normalizing IGF-I levels in treatment naive patients with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acromegaly
* IGF-I levels >=1.3xULN (upper limit of normal) at screening
* No history of radiotherapy or prior treatment with other drugs for acromegaly
* Minimum of two months must have elapsed post surgery prior to screening

Exclusion Criteria:

* Presence of other conditions that may result in abnormal GH (Growth Hormone) and/or IGF-I concentrations
* AST/ALT >= 3xULN (upper limit of normal)
* Pituitary adenoma within 3mm of optic chiasm confirmed by recent MRI
* Visual field defects (except post surgical stable residual defects)
* Unable to self administer drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-04; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with normal IGF-1 concentration at Final Visit (Week 52)

SECONDARY OUTCOMES:
The secondary endpoints include: 1.Percentage of patients with normal IGF-I concentration at any visit. 2.Percent change from Baseline of IGF-I at each visit. 3.Percent change from Baseline of IGFBP-3 (IGF binding protein-3) at Week 24 and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (11):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
- Australia (4):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Fitzroy, Victoria
  - Pfizer Investigational Site, Heidelberg, Victoria
- Brazil (4):
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (3):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Montreal, Quebec
- France (2):
  - Pfizer Investigational Site, Le Kremlin-Bicêtre
  - Pfizer Investigational Site, Pessac
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Marburg
- Greece (2):
  - Pfizer Investigational Site, Athens, Attika/Greece
  - Pfizer Investigational Site, Piraeus
- Ireland (2):
  - Pfizer Investigational Site, Cork
  - Pfizer Investigational Site, Dublin
- Italy (5):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Torino
- Pfizer Investigational Site, Oslo, Norway
- Spain (4):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
- Sweden (4):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- United Kingdom (3):
  - Pfizer Investigational Site, Belfast, Ireland
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=PEGA-0435-003&StudyName=A+Study+To+Compare+The+Efficacy+And+Safety+Of+Pegvisomant+To+That+Of+Sandostatin+Lar+Depot+In+Patients+With+Acromegaly